CLINICAL TRIAL: NCT02469805
Title: Stimulated Versus Un-stimulated Intrauterine Insemination Cycles in Couples With Mild Male Factor Infertility: A Randomized Controlled Trial
Brief Title: Stimulated Versus Un-stimulated Intrauterine Insemination Cycles in Couples With Mild Male Factor Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sub 12
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — hMG-IBSA; Ovulation Detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- stimulated intrauterine insemination (IUI) (Active Comparator): On the 3rd day of menstruation women in group 1 will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins starting from the 3rd day of menstruation. On day 8 the ultrasound will be repeated and serum E2 will be measured, hMG dose will be adjusted and continued and the frequency of ultrasound scans will be individualized. HMG will be stopped when at least 2 follicles measuring 18 mm are associated with serum E2 of 500-3000 Pg/mL, this was followed by the administration of 10000 IU of human chorionic gonadotropin
  Interventions: Drug: Merional; Drug: Choriomon; Procedure: IUI; Device: Shepherd catheter
- Unstimulated IUI (Active Comparator): Women in group 2 will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit. IUI will be performed on the day after the surge in urinary excretion of luteinizing hormone.
  Interventions: Procedure: IUI; Procedure: Ovulation detection; Device: Shepherd catheter
- Control group (Active Comparator): Women will be asked to test their urine for luteinizing hormone by the same method as group 2. They will be asked to have an intercourse on the day after the surge in urinary excretion of luteinizing hormone and this will be repeated for 12 months.
  Interventions: Procedure: Ovulation detection

INTERVENTIONS:
Drug: Merional — On the 3rd day of menstruation women will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins (hMG, Merional ®, IBSA, Lugano, Switzerland) starting from the 3nd day of menstruation.
  Arms: stimulated intrauterine insemination (IUI)
Drug: Choriomon — Administration of 10000 IU of human chorionic gonadotropin (hCG; Choriomon®, IBSA) when at least 2 follicles measuring 18 mm are observed during vaginal ultrasound and is associated with serum E2 of 500-3000 Pg/mL.
  Arms: stimulated intrauterine insemination (IUI)
Procedure: IUI — Semen will be processed and drawn into a shepherd catheter attached to a 1 mL syringe and injected into the uterus
  Arms: Unstimulated IUI; stimulated intrauterine insemination (IUI)
Procedure: Ovulation detection — Women will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit
  Arms: Control group; Unstimulated IUI
Device: Shepherd catheter — Processes semen will be drawn into a shepherd catheter attached to a 1 mL syringe and injected into the uterus
  Arms: Unstimulated IUI; stimulated intrauterine insemination (IUI)

SUMMARY:
Four hundred and fifty women with mild male factor infertility will be divided into 3 equal groups using computer generated random numbers: Group 1 will have up to 4 stimulated IUI cycles, group 2 will have up to 4 unstimulated cycles, women who do not become pregnant after the 4 cycles in groups 1 and 2 will be advised to have regular intercourse at the expected time of ovulation. Group 3 will be the control group will be advised to have regular sexual intercourse at the time of ovulation for 6 months

DETAILED DESCRIPTION:
Mild male factor infertility is defined as: Two or more semen analyses that have one or more variables which fall below the 5th centile as defined by the World Health Organization, and where the effect on the chance of pregnancy occurring naturally through vaginal intercourse within a period of 24 months would then be similar to people with unexplained infertility or mild endometriosis. The application of ovarian stimulation in IUI is advocated, even if the woman has ovulatory cycles, to improve the pregnancy rates with IUI. However, the application of ovarian stimulation has two main drawbacks: The increased chances of a multiple pregnancy and ovarian hyperstimulation syndrome. To avoid these complications unstimulated IUI cycles have been investigated. The objective of the study is to evaluate the role of stimulated and unstimulated IUI cycles in the management of mild male factor infertility.

The study will be conducted in Cairo university hospitals and BeniSuef University hospitals All patients with mild male factor infertility attending both sites will be invited to participate in the study. The study will be explained and only couples who sign written consents will be included in the study.

Four hundred and fifty women with mild male factor infertility will be divided into 3 equal groups using computer generated random numbers: Group 1 will have up to 4 stimulated IUI cycles, group 2 will have up to 4 unstimulated cycles, women who do not become pregnant after the 4 cycles in groups 1 and 2 will be advised to have regular intercourse at the expected time of ovulation. Group 3 will be the control group will be advised to have regular sexual intercourse at the time of ovulation for 6 months On the 3rd day of menstruation group 1 will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins (hMG, Merional ®, IBSA, Lugano, Switzerland) starting from the 3nd day of menstruation. On day 8 the ultrasound will be repeated and serum E2 will be measured, hMG dose will be adjusted and continued and the frequency of ultrasound scans will be individualized. HMG will be stopped when at least 2 follicles measuring 18 mm are associated with serum E2 of 500-3000 Pg/mL, this was followed by the administration of 10000 IU of human chorionic gonadotropin (hCG; Choriomon®, IBSA) Women in group 2 will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit. Intrauterine insemination will be performed on the day after the surge in urinary excretion of luteinizing hormone.

Women in group 3 will be asked to test their urine for luteinizing hormone by the same method as group 2. They will be asked to have an intercourse on the day after the surge in urinary excretion of luteinizing hormone and this will be repeated for 12 months.

Semen specimens for groups 1 and 2 will be evaluated and prepared for IUI within one hour after collection. Semen will be diluted 1:2 (vol/vol) with HEPES-buffered Ham's F10 medium containing 1.5 percent serum albumin. After centrifugation for 10 minutes, the pellets will be re-suspended and combined in 3 ml of the medium.

The sperm suspension will be centrifuged for 10 minutes, and the pellet was resuspended in 0.35 ml of medium. Approximately 0.05 ml will be used to determine the concentration and motility of sperms. The remaining sample will be drawn into a shepherd catheter attached to a 1 mL syringe and injected into the uterus.

The procedure will be repeated for up to 4 months in groups 1 and 2, if pregnancy does not occur. Women who do not conceive after the 4 trials will be asked to check their urine for luteinizing hormone using the ovulation detection kits and have an intercourse on the day following the luteinizing hormone surge. This will be repeated for 8 months.

The pregnancy rates of the 3 groups will be compared after the 4 months and after one year.

ELIGIBILITY:
Inclusion Criteria:

* Mild male factor infertility defined as meaning two or more semen analyses that have one or more variables which fall below the 5th centile as defined by the World Health Organization, and where the effect on the chance of pregnancy occurring naturally through vaginal intercourse within a period of 24 months would then be similar to people with unexplained infertility or mild endometriosis.

Exclusion Criteria:

* Known allergy to FSH
* Other factors of infertility.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after IUI or timed sexual intercourse

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HW, Behre HM, Haugen TB, Kruger T, Wang C, Mbizvo MT, Vogelsong KM. World Health Organization reference values for human semen characteristics. Hum Reprod Update. 2010 May-Jun;16(3):231-45. doi: 10.1093/humupd/dmp048. Epub 2009 Nov 24. PMID 19934213
- [Background] Quintero RB, Urban R, Lathi RB, Westphal LM, Dahan MH. A comparison of letrozole to gonadotropins for ovulation induction, in subjects who failed to conceive with clomiphene citrate. Fertil Steril. 2007 Oct;88(4):879-85. doi: 10.1016/j.fertnstert.2006.11.166. PMID 17920403